CLINICAL TRIAL: NCT03860623
Title: The Effect of Oral Feeding on Gastric Emptying, Small Bowel Water Content, Superior Mesenteric Artery Blood Flow, Plasma Hormone Concentrations and Blood Volume in Obese and Healthy Weight Subjects.
Brief Title: Effect of Oral Feeding on Gastric Emptying, Gut Blood Flow, and Hormone Responses in Obese and Healthy Weight Subjects
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Elizabeth Simpson, Senior Research Fellow, University of Nottingham
Other Study IDs: A16042015
Record Dates: First submitted 2019-02-25; First posted 2019-03-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Obesity
Keywords: satiety; gut blood flow; gastric emptying; obesity; incretin hormones
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Overweight: Otherwise healthy overweight and obese men (BMI 30-40kg/m2) aged 18 to 60 years Group will consume a standard meal (Feeding) and measurements will be made before (baseline) and for 300 minutes after eating
- Normal Weight: Healthy normal weight men (BMI 18-25kg/m2, but including those with BMI up to 28kg/m2 if waist circumference <96cm) aged 18 to 60 years Group will consume a standard meal (Feeding) and measurements will be made before (baseline) and for 300 minutes after eating

SUMMARY:
Obesity is a complicated condition that is poorly understood. The aim of this study is to increase our knowledge of how the condition may arise, and what makes obese people remain obese.

We will be investigating 12 people who are overweight and comparing them to 12 people who are lean, to look at how quickly food empties out of the stomach (gastric emptying) and travels through the gut, what the blood flow to the gut is, and also to examine the hormones which are involved in determining how full people feel after eating. In order to do this, we will be using a magnetic resonance imaging (MRI) scanner, and performing blood tests.

The rate of gastric emptying may have an impact on satiety (how full one feels) and has been implied in the development of obesity. This effect has been shown to impact on subsequent meal intake to a greater degree in overweight subjects, and may be due to a difference in gastric emptying of food in overweight individuals, or to hormones such as ghrelin, glucagon-like peptide 1, and Peptide YY.

DETAILED DESCRIPTION:
The World Health Organisation (WHO) has deemed being overweight or obese as the fifth leading cause for global deaths, with more than 1.9 billion adults being defined as overweight, and 600 million defined as being obese. Conditions associated with obesity, such as stroke, type 2 diabetes, certain cancers, cardiovascular, fatty liver and airway disease can lead to premature death. Obesity results from an imbalance in energy intake versus expenditure, and fat mass accumulates. Studies have indicated that obese animals have a faster gastric emptying time, a weaker contraction of the duodenum, but a stronger contraction and relaxation of the ileum, with associated changes in gastrointestinal neurohormonal levels. The rate of gastric emptying may have an impact on feelings of satiety and has been implied in the pathogenesis of obesity. Moreover, mesenteric blood flow increases 3-fold following a meal and in a swine experimental model, a reduction in weight gain was seen when blood flow was intentionally limited to the gut using flow-restricting endovascular stenting. The authors concluded that this intervention may play a role in the treatment of obesity where other interventions have failed or are inappropriate; however the role of blood flow to the gut in obese individuals is important to elucidate. We hypothesize that nutrient absorption in obese and healthy weight individuals after a standardized meal is determined by differences in gastric emptying and mesenteric blood flow which give rise to different insulin, glucose and gut hormone responses. These may be contributory mechanisms to the evolution or maintenance of obesity.

The aim of this study is to establish the effects of food ingestion on gastric emptying, gallbladder emptying, small bowel water content and splanchnic blood flow as measured by serial magnetic resonance imaging (MRI) in the context of changes in plasma gastrointestinal hormone secretion in human subjects who are obese or healthy weight. In addition, this pilot study will provide the data necessary to power a larger study investigating methods of dietary manipulation in the treatment of obesity.

Method: In order to normalize the pre-study diet, volunteers will have consumed a standard diet for the 3 days immediately before the study visit, which will be based on foods in their normal diet and will be designed to meet their estimated energy requirements and provide 15% of total daily energy intake as protein, 35% as fat and 50% as carbohydrate. Participants will report at 0800 hours following a fast from midnight and after having abstained from alcohol, nicotine, and caffeine from 1800 hours the day before. On arrival, participants will be given a drink of water (200ml). A retrograde cannula will be inserted into a dorsal foot vein after prior intradermal infiltration of 1% lidocaine, with the foot placed in a magnetic resonance (MR) compatible warming box that we have developed, for arterialized-venous blood sampling. Prior to baseline blood sampling, participants will undergo a magnetic resonance imaging (MRI) scan to determine baseline values for superior mesenteric artery (SMA) blood flow, small bowel water content and gastric fluid and gas volumes. Liver fat, visceral fat and subcutaneous fat volumes will also be assessed at this time. Subsequently, a blood sample will be drawn for analysis of concentrations of hemoglobin, glucose, insulin, glucagon-like peptide 1 (GLP-1), glucagon-like peptide 2 (GLP-2), ghrelin and peptide YY (PYY). Serum osmolality will also be measured and subjective appetite assessed using visual analogue scales. The participants will then be given the test meal (in an upright, seated position) and asked to consume it within 15 minutes. The test meal will be comprised of pasta, cheese and tomato sauce, and provides 13% of total energy (E) from protein, 39%E fat, and 48%E carbohydrate.

Following the test meal (time = 0 minutes), subjective appetite will be measured as before, then participants will be scanned at 30 minute intervals for 4 hours to assess gastric emptying, gastric accommodation, gastric motility and small bowel water content, as well as SMA blood flow. Blood samples will be drawn at 15 minutes, then every half hour until 240 minutes after the test meal, with a final blood sample taken at 300 minutes. Subjective appetite will be assessed every hour over the 300 minute study.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-40 kg/m2
* BMI 18-25 kg/m2; those with BMI up to 28kg/m2 will be included if waist circumference is <96cm.
* Males
* Aged 18-60yrs

Exclusion Criteria:

* Acute illness in the preceding 6 weeks
* Taking regular medication
* History of deep vein thrombosis or clotting disorders
* Hypertension
* Diabetes
* Any clinically significant findings at screening
* History of substance abuse
* Demonstrating factors precluding safe MRI
* History of gastrointestinal motility disorders (e.g. gastroesophageal reflux disease -irritable bowel syndrome, gastroparesis, sphincter of Oddi dysfunction, etc.)
* Previous thoracic or abdominal surgery.
* Those who report having ≤3 bowel movements/week or >2/day.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recruitment will be from the male population residing within 20 miles of the research site. This will include those from Nottinghamshire, Leicestershire and Derbyshire, UK
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Gastric emptying rate | 240 minutes after feeding
  time taken for a standard meal to empty from the stomach, assessed by serial volume measurements of the stomach using magnetic resonance imaging

SECONDARY OUTCOMES:
Stomach volume in the fasted state | baseline
  volume of the stomach measured by magnetic resonance imaging
Superior mesenteric artery (SMA) blood flow in the fasted state | baseline
  blood flow in the SMA assessed using magnetic resonance imaging
superior mesenteric artery (SMA) blood flow response to feeding | 240 minutes after feeding
  blood flow response to feeding, determined in the SMA every half hour using magnetic resonance imaging
Fasting blood glucose concentration | before feeding
  whole blood glucose concentration assessed using a Hemocue glucose analyser
Blood glucose response to feeding | 300 minutes after feeding
  whole blood glucose concentration response to feeding, assessed by serial sampling using a Hemocue glucose analyser
Fasting insulin concentration | baseline
  serum insulin concentration in the fasted state measured at a later date using a radio-immunoassay (RIA)
serum insulin response to feeding | 300 minutes after feeding
  serum insulin concentration response to feeding, assessed by serial sampling and measured at a later date using a RIA
Fasting plasma GLP-1 concentration | baseline
  Plasma GLP-1 concentration in the fasted state, measured at a later date using an enzyme-linked immunosorbent assay (ELISA)
Plasma GLP-1 response to feeding | 300 minutes after feeding
  Plasma GLP-1 concentration response to feeding, assessed by serial sampling and measured at a later date using an ELISA
Fasting plasma GLP-2 concentration | baseline
  Plasma GLP-2 concentration in the fasted state, measured at a later date using an enzyme-linked immunosorbent assay (ELISA)
Plasma GLP-2 response to feeding | 300 minutes after feeding
  Plasma GLP-2 concentration response to feeding, assessed by serial sampling and measured at a later date using an ELISA
Fasting plasma Ghrelin | baseline
  Plasma Ghrelin concentration in the fasted state measured at a later date using a RIA
Plasma Ghrelin response to feeding | 300 minutes after feeding
  Plasma Ghrelin concentration response to feeding assessed by serial sampling and measured at a later date using a RIA
Fasting plasma peptide YY (PYY) | baseline
  Plasma PYY concentration in the fasted state measured at a later date using a RIA
Plasma peptide YY (PYY) response to feeding | 300 minutes after feeding
  Plasma PYY concentration response to feeding assessed by serial sampling and measured at a later date using a RIA
Subjective satiety in the fasted state | baseline
  Satiety of individuals in the fasted state will be assessed using 4 visual analogue scales ('How hungry do you feel', 'how much food do you think that you could eat', how strong is your desire to eat' and how full do you feel')
Subjective satiety after eating | immediately after eating the standard meal
  Satiety immediately after eating the standard meal will be assessed using 4 visual analogue scales ('How hungry do you feel', 'how much food do you think that you could eat', how strong is your desire to eat' and 'how full do you feel')
Subjective satiety response to eating | 300 minutes after eating
  The satiety response to the standard meal will be assessed over the 300 minute study period using hourly collection of 4 visual analogue scales ('How hungry do you feel', 'how much food do you think that you could eat', how strong is your desire to eat' and 'how full do you feel')
visceral adiposity | baseline
  amount of visceral fat present, determined by MRI of the torso
subcutaneous adiposity | before feeding
  thickness of the subcutaneous fat layer on the torso, determined by MRI
hepatic lipid content | baseline
  liver triacylglyceride content will be estimated using proton magnetic resonance spectroscopy
Attrition rate | 1 year
  Number of participants completing the protocol as a proportion of those who were recruited to the study
Recruitment rate | 1 year
  number of people volunteering to take part in the study as a proportion of those expressing initial interest

CONTACTS AND LOCATIONS:
Overall Officials: Dileep Lobo, MD, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Queens Medical Centre, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu XY, Li Z, Zhang N, Yu HT, Wang SR, Liu JR. Effects of gastrointestinal motility on obesity. Nutr Metab (Lond). 2014 Jan 7;11(1):3. doi: 10.1186/1743-7075-11-3. PMID 24398016
- [Background] Vatner SF, Franklin D, Van Citters RL. Mesenteric vasoactivity associated with eating and digestion in the conscious dog. Am J Physiol. 1970 Jul;219(1):170-4. doi: 10.1152/ajplegacy.1970.219.1.170. No abstract available. PMID 4393203
- [Background] Alyami J, Spiller RC, Marciani L. Magnetic resonance imaging to evaluate gastrointestinal function. Neurogastroenterol Motil. 2015 Dec;27(12):1687-92. doi: 10.1111/nmo.12726. PMID 26598049
- [Background] Hoad CL, Parker H, Hudders N, Costigan C, Cox EF, Perkins AC, Blackshaw PE, Marciani L, Spiller RC, Fox MR, Gowland PA. Measurement of gastric meal and secretion volumes using magnetic resonance imaging. Phys Med Biol. 2015 Feb 7;60(3):1367-83. doi: 10.1088/0031-9155/60/3/1367. Epub 2015 Jan 16. PMID 25592405
- [Background] Totman JJ, Marciani L, Foley S, Campbell E, Hoad CL, Macdonald IA, Spiller RC, Gowland PA. Characterization of the time course of the superior mesenteric, abdominal aorta, internal carotid and vertebral arteries blood flow response to the oral glucose challenge test using magnetic resonance imaging. Physiol Meas. 2009 Oct;30(10):1117-36. doi: 10.1088/0967-3334/30/10/011. Epub 2009 Sep 16. PMID 19759401
- [Result] Simpson EJ, Althubeati S, Cordon S, Hoad C, Bush D, Eldeghaidy S, Gowland PA, Macdonald IA, Lobo DN. The effect of oral feeding on gastrointestinal function, motility and appetite-regulating hormones, insulin, glucose and satiety in normal weight individuals and those with obesity. Clin Nutr. 2025 Sep;52:62-71. doi: 10.1016/j.clnu.2025.07.008. Epub 2025 Jul 8. PMID 40714600
- See also: WHO estimation of Global Overweight and Obesity — http://www.who.int/mediacentre/factsheets/fs311/en/.